CLINICAL TRIAL: NCT05938452
Title: A Phase 1, Randomized, Double-Blind, Single-Dose Escalation Study Followed by a Multiple-Dose Escalating Study of Glyceryl Tribenzoate (GTB) Capsules in Healthy Subjects
Brief Title: Safety and Tolerability of Glyceryl Tribenzoate (GTB) Capsules in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Forest Hills Lab (Industry)
Collaborators: Liberyx Therapeutics Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FHL-101-001
Record Dates: First submitted 2023-06-15; First posted 2023-07-10 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2023-06

CONDITIONS: Neurological Disorder
MeSH Terms: conditions — Nervous System Diseases | interventions — glyceryl tribenzoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Active Comparator
  Interventions: Drug: Glyceryl Tribenzoate
- Placebo (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Glyceryl Tribenzoate

INTERVENTIONS:
Drug: Glyceryl Tribenzoate — Oral Solution

SUMMARY:
This study is designed to assess the safety and PK/PD of GTB and Benzoic Acid (Benzoate) using a single ascending dose (SAD) study (under fasting conditions).

DETAILED DESCRIPTION:
This study is designed to assess the safety and PK/PD of GTB and Benzoic Acid (Benzoate) using a single ascending dose (SAD) study (under fasting conditions). After a wash out period, a cohort under fed conditions (ingestion of a high-fat morning meal) will be evaluated. Following the SAD, the multiple ascending dose phase will take place with two different cohorts. A battery of labs, hematology, physical examinations including vital signs, and ECGs will be monitored throughout the study for assessment of the study drug (GTB) compared with placebo. The clinical and laboratory data (excluding PK/PD data) of each cohort will be evaluated by a Data Monitoring Committee (DMC) to allow escalation to the next dose level during the SAD and MAD portions of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to any study-related procedures.
2. Male or female subjects 18 to 50 years of age inclusive.
3. Subject's body mass index (BMI) is ≥ 18 kg/m2 and ≤ 30 kg/m2.
4. Female subjects of childbearing potential must not be pregnant or lactating with a negative serum human chorionic gonadotropin (HCG) pregnancy test result at Screening, and negative urine pregnancy test on Day -1 (including Day -1 of Period 2 for SAD dosing participants i.e., fed cohort).
5. Female subjects of childbearing potential must use an adequate method of contraception from Screening until 30 days after last dose of study medication. Acceptable methods of contraception are barrier methods (female condom, diaphragm, cervical cap, spermicide, or intrauterine device [IUD]), surgical sterility (self-reported: tubal ligation, hysterectomy, and/or bilateral oophorectomy), oral hormonal contraceptives, hormonal IUD, and/or postmenopausal status (defined as at least 1 year without menses as demonstrated by medical history or subject report).
6. Male subjects must use an adequate method of contraception from Screening until 30 days after last dose of study medication. Acceptable methods of contraception are barrier methods (condom), surgical sterility (self-reported), must also refrain from donating sperm while on study medication and until 30 days after last dose of study medication.
7. Subject is in good health as determined by vital signs, medical history, physical exam, ECG, and safety laboratory analyses at Screening and during the study.
8. Subject is negative for SARS-CoV-2 virus at admission Day -1 and Day 1 (during the SAD, Fed portion of the study, and MAD).
9. Subject does not have dysphagia and discomfort with swallowing tablets/capsules.

Exclusion Criteria:

1. Subject has used an investigational product or device within 30 days prior to enrollment or during the study.
2. Subject has used prescription or non-prescription drugs (including vitamins, minerals, and herbal/plant-derived preparations) within 2 weeks of enrollment (excluding hormonal IUD, oral hormonal contraceptives, hormone replacement therapy, and acetaminophen) unless deemed acceptable by the Investigator in consultation with the Sponsor.
3. Subject has a positive drug and/or alcohol test at Screening and on Day -1 (including 4. Day -1 of Period 2 for SAD dosing participants, i.e., fed cohort).
4. Subject has a history of drug or alcohol abuse within 2 years before Screening.
5. Subject is unable to abstain from ingesting alcohol or smoking for 72 hours prior to dosing and throughout the study.
6. Concurrent use of probenecid, penicillin or other ß-lactams, or other drugs which undergo active tubular secretion in the kidneys.
7. The subject has a clinically significant history of endocrinologic, hematologic, hepatic, immunologic, metabolic, cardiovascular, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major diseases or malignancy.
8. Allergy to sodium benzoate.
9. Has an active suicidal plan/intent or have had active suicidal thoughts in the past 6 months or a suicide attempt in the past 3 years.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events | 7 days
  Incidence of Treatment-Emergent Adverse Events (TEAEs) until 30 days after the last administration of the study medication.
  6. Change from baseline in 12-lead electrocardiogram (ECG).
Treatment-Emergent Adverse Events Withdrawals | 7 days
  Incidence of TEAEs leading to withdrawal of study drug or study discontinuation.
Laboratory Results | 7 days
  Change from baseline in clinical laboratory results.
Physical Results | 7 days
  Change from baseline in physical examination results
Vital Signs | 7 days
  Change from baseline in vital signs.
Electrocardiogram | 7 days
  Change from baseline in 12-lead electrocardiogram (ECG).

CONTACTS AND LOCATIONS:
Locations (1):
- TKL Research, Bloomfield, New Jersey, United States